CLINICAL TRIAL: NCT03399357
Title: Evaluation of Metabolic Predictors of Influenza Vaccine Immune Response in the Singapore Elderly Population- the DYNAMIC Trial
Brief Title: Evaluation of Metabolic Predictors of Influenza Vaccine Immune Response in the Singapore Elderly Population - the DYNAMIC Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Singapore Immunology Network (Unknown); National Healthcare Group, Singapore (Other Government)
Responsible Party: Sponsor
Other Study IDs: DSRB 2016/00248
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Influenza Vaccine; Immune Response; Elderly; Vitamin D Deficiency; Metabolic Disease; Diabetes Mellitus
MeSH Terms: conditions — Influenza, Human; Vitamin D Deficiency; Metabolic Diseases; Diabetes Mellitus | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood samples at "baseline" i.e. Day 0 to D -7 from Vaccination Day (designated as Day 0) and Day 28 +/- 3 post-vaccination to assess HAI (hemagglutinin inhibition) response.
     PBMCs to be stored for future studies.
  2. Baseline blood sample to be tested for 25-OH D assay.
  3. Stool samples (optional part of study) to be studied for stool microbiome and relation to immune response and Vitamin D status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ≥ 65 Years old: Healthy community-dwelling elderly (men and women) age 65 and above who are eligible for influenza vaccine and fulfil inclusion and exclusion criteria
  Interventions: Biological: Influenza Vaccine

INTERVENTIONS:
Biological: Influenza Vaccine — Inactivated Trivalent Influenza Vaccine (IIV3) 2017 containing: A (H1N1): an A/Michigan/45/2015 (H1N1) - like virus (new strain); A (H3N2): an A/Hong Kong/4801/2014 (H3N2) - like virus; B/Brisbane/60/2008 - like virus
  Other Names: Influvac(R) SH 2017

SUMMARY:
The trial aims to evaluate role of metabolic factors including systemic 25-OH D and diabetes in the adaptive immune response (haemagluttination inhibition titer) to influenza vaccine in the elderly. The influenza vaccine administered in this study will be licensed trivalent inactivated influenza vaccine. Elderly who are age above 65 including those with co-morbidities such as diabetes mellitus will be included. The study has its inclusion and exclusion criteria to determine eligibility for participation.

DETAILED DESCRIPTION:
Novel, effective influenza vaccination strategies are needed in the elderly who have the highest rate of influenza-related morbidity and mortality. Vaccine efficacy in the elderly is reduced due to immunosenescence and/or, inflamm-aging. This phase IV clinical trial in 240 participants aims to evaluate metabolic predictors of influenza-vaccine specific immune response in a multi-ethnic elderly community cohort in Singapore. Specifically, our novel approach is to evaluate the immunomodulatory roles of vitamin D, diabetes and other metabolic predictors. This study has translational implications (e.g. using vitamin D as an 'adjuvant', evaluating biomarkers of vaccine efficacy) to enhance influenza vaccine immunogenicity in the vulnerable elderly.

Potential benefit: there is a possibility the vaccine may prevent influenza illness or influenza related complication that might have otherwise occurred. This study will contribute to body of knowledge of impact of metabolic factors (vitamin D, DM status) on influenza vaccine immune response, and will be the first study of its kind to be done in an Asian elderly population. Potential risks related to the blood draw and local/systemic side effects from influenza vaccine are anticipated to be minimal.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and above at time of enrollment (up to age 100) and able to give informed consent
* Determined by medical history, physical examination, and clinical judgment to be generally healthy, with no immunosuppressive conditions and having stable current medical conditions. Subjects with preexisting, stable disease, defined as not requiring significant change in therapy or hospitalization for worsening of disease 12 weeks prior to receipt of study vaccine are eligible. A change in dose or therapy within a treatment category (e.g., change from one non-steroidal anti-inflammatory drug to another) is allowed. A change to a new therapy category (e.g., surgery or addition of a new pharmacological class) is only allowed if it is not caused by worsening disease.
* Is eligible for seasonal influenza vaccine
* Is available for all planned study visits
* Is willing to follow study procedures
* Able to follow study procedures (questionnaires, blood draws, vaccination) in the opinion of the investigator

Exclusion Criteria:

* A change to a new therapy category caused by worsening disease is considered significant and will disqualify subject from participating in the study
* Subjects reporting any symptoms suggestive of influenza, influenza-like illness, or respiratory illness
* Vaccination with any licensed or experimental influenza vaccine within the past 10 months
* Intent to receive any other investigational vaccine or agent during the course of the study
* Intent to receive other licensed vaccines during the course of the study (does not apply for pandemic or post-exposure prophylaxis scenario
* History of severe adverse reaction associated with an influenza vaccine
* Allergic to egg proteins (egg or egg products) and chicken proteins
* Known or suspected immunodeficiency or receiving treatment with immunosuppressive therapy including cytotoxic agents in past 6 months e.g., transplant recipients on active immunosuppression, patients with cancer, HIV, or autoimmune disease.
* Long-term systemic corticosteroid therapy (prednisolone ≥ 7.5mg/day or equivalent for more than 2 consecutive weeks within the past 3 months) Note: If systemic corticosteroids have been administered short term for treatment of an acute illness, subjects will be excluded from the study until corticosteroid therapy had been discontinued for at least 30 days.
* History of Guillain-Barré syndrome
* Serious chronic medical condition including: metastatic malignancy, severe chronic obstructive pulmonary disease requiring supplemental oxygen, CKD stage 3 and above, end stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that in the investigator's opinion should preclude the subject from participating in the study
* Bariatric surgery, GI malabsorption disorders
* Recurrent Falls (≥2 falls in the past 12 months)
* Osteoporosis with or without pathological fractures
* Current or recently completed high dose vitamin D supplementation within the past 3 months (defined as daily cholecalciferol dose of 2000 IU or higher, weekly 50,000 IU or intramuscular calcitriol)
* Receipt of any blood products, including immunoglobulin, within six months of study enrollment
* Donated blood within last 58 days
* Current anticoagulant therapy or a history of bleeding diathesis (including thrombocytopenia with platelet count < 50,000) that would contraindicate intramuscular (IM) injection (Note: antiplatelet drugs such as aspirin and clopidogrel are permitted)
* Moderate or severe acute illness/infection (according to investigator judgement) on the day of vaccination, or febrile illness (temperature ≥ 37.5°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided.
* Any medical condition that would, in the opinion of the investigator, interfere with the evaluation of the study objectives

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy elderly population with stable comorbidities (in particular diabetes mellitus) is chosen for this study to evaluate metabolic factors and predictors related to immunosenescence, inflamm-aging and immune response to vaccination. Vaccination is one of our key preventive measures for influenza yet additional insight is needed regarding adaptive response in this vulnerable population, to ultimately lead to novel vaccination strategies.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Humoral immune response measure | Day 0 to Day 28 post vaccination
  Haemagglutination inhibition (HAI) titer for each of the three influenza vaccine strains in response to influenza vaccine at day 28 compared to baseline (pre-vaccination) titer

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No